CLINICAL TRIAL: NCT01354639
Title: Comparative Study of Surgical Completeness After Robotic Thyroidectomy Versus Conventional Open Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0082
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Group 1 : conventional open thyroidectomy group (papillary thyroid carcinoma patient who underwent conventional open bilateral total thyroidectomy procedure and postoperative low dose RAI therapy)
- Group 2: Group 2 : robotic thyroidectomy group (papillary thyroid carcinoma patient who underwent robotic bilateral total thyroidectomy procedure and postoperative low dose RAI therapy)

SUMMARY:
The robotic thyroidectomy (RT) has excellent cosmetic and several functional results. But there were no definite evidence of oncological safety of robotic thyroidectomy yet. To assure the surgical completeness of robotic thyroidectomy, the investigators compared robotic thyroidectomy and conventional open thyroidectomy (OT) by means of the postoperative radioactive iodine (RAI) uptake of possible remnant thyroid tissue and stimulated TG level.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20years
* papillary thyroid carcinoma patients who underwent conventional open or robotic bilateral total thyroidectomy at YUHS(Yonsei University Health System)
* patient who underwent postoperative low doe (30mCI) RAI ablation therapy at YUHS

Exclusion Criteria:

* pregnant, lactating women
* patient who underwent postoperative low dose RAI at another hospital
* patient with distant metastasis
* patient who underwent combined operation with bilateral total thyroidectomy (ex) Modified radical neck dissection, selective neck node excision d/t lateral neck node metastasis
* patient who underwent High dose (more than 30 mCI) RAI therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: papillary thyroid carcinoma patient who underwent conventional open or robotic bilateral total thyroidectomy procedure and postoperative low dose RAI therapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
surgical completeness of conventional open thyroidectomy and robotic thyroidectomy | 12 months after low dose RAI albation therapy
  check remnant thyroid uptake at Diagnostic RAI scan and stimulated serum thyroglobulin level

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kang SW, Lee SC, Lee SH, Lee KY, Jeong JJ, Lee YS, Nam KH, Chang HS, Chung WY, Park CS. Robotic thyroid surgery using a gasless, transaxillary approach and the da Vinci S system: the operative outcomes of 338 consecutive patients. Surgery. 2009 Dec;146(6):1048-55. doi: 10.1016/j.surg.2009.09.007. Epub 2009 Oct 30. PMID 19879615
- [Background] Kang SW, Jeong JJ, Nam KH, Chang HS, Chung WY, Park CS. Robot-assisted endoscopic thyroidectomy for thyroid malignancies using a gasless transaxillary approach. J Am Coll Surg. 2009 Aug;209(2):e1-7. doi: 10.1016/j.jamcollsurg.2009.05.003. Epub 2009 Jun 12. No abstract available. PMID 19632588
- [Background] Kang SW, Jeong JJ, Yun JS, Sung TY, Lee SC, Lee YS, Nam KH, Chang HS, Chung WY, Park CS. Robot-assisted endoscopic surgery for thyroid cancer: experience with the first 100 patients. Surg Endosc. 2009 Nov;23(11):2399-406. doi: 10.1007/s00464-009-0366-x. Epub 2009 Mar 5. PMID 19263137
- [Background] Lee J, Nah KY, Kim RM, Ahn YH, Soh EY, Chung WY. Differences in postoperative outcomes, function, and cosmesis: open versus robotic thyroidectomy. Surg Endosc. 2010 Dec;24(12):3186-94. doi: 10.1007/s00464-010-1113-z. Epub 2010 May 19. PMID 20490558